CLINICAL TRIAL: NCT04916977
Title: Global Burden and Treatment Trajectiories in Italian Patients With Fabry Disease: a Retrospective, Longitudinal and Cross-sectional Study
Brief Title: Global Burden and Treatment Trajectiories in Italian Patients With Fabry Disease
Acronym: GROUND
Status: Completed | Type: Observational
Sponsor: Chiesi Italia (Industry)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Other Study IDs: DFIDM-2001
Record Dates: First submitted 2021-05-13; First posted 2021-06-08 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; Rare; Retrospective; Burden
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FD patients
  Interventions: Other: FD patients

INTERVENTIONS:
Other: FD patients — Patients with Fabry disease diagnosis

SUMMARY:
GROUND study is an Italian, multicenter retrospective longitudinal cohort study with a cross-sectional phase with the aim to quantify the severe clinical burden in terms of severe and fatal outcomes and extension of clinical impairment in the Italian Fabry Disease patients' population

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients living or deceased of either sex (age ≥18 years) with a documented FD diagnosis in the last 10 years from the beginning of the study.
2. Patients with at least 3 years of follow-up or early occurrence of severe/fatal outcomes. Also, adult patients who were lost by their care provider or physician and cannot be traced, but for which it is possible to retrieve data for at least 3 years before the last available follow-up visit or from diagnosis to the occurrence of severe/fatal outcomes if earlier, can be included.
3. Written informed consent to undergo in the cross-sectional protocol clinical visit and to retrospectively collect genetic/clinical data. In case of deceased or untraceable patients, the written informed consent is not required to collect retrospective clinical data (excluding genetic data).

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed FD diagnosis
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of severe and fatal clinical outcomes | Baseline
  Occurrence of severe and fatal clinical outcomes derived by event-free survival from birth to last follow-up or cross-sectional visit;
Comprehensive burden | Baseline
  Comprehensive burden intended as a measure of extension of clinical impairment assessed by median Mainz Severity Score Index (MSSI) at last follow-up or cross-sectional visit.

SECONDARY OUTCOMES:
Percentage of patients with disease progression | From the first available FASTEX score to baseline
  Percentage of patients with disease progression measured by FAbry STabilization indEX and defined as a change >20% from the first available FASTEX score to the last follow-up and in the last 2 years until the last follow-up and 2 years before the last follow-up or cross-sectional visit (or when available within 3-1 years before last follow-up)
Percentage of patients with disease activity | Baseline
  Percentage of patients with disease activity assessed by the occurrence rate of clinically significant events from diagnosis to last follow-up or cross-sectional visit.
Brief pain inventory score | Baseline
  Uses simple numeric rating scales from 0 (no pain) to 10 (severe pain)
Pittsburgh Sleep Quality index | Baseline
  Seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Hamilton depression scale | Baseline
  It contains 17 items. A score of 0-7 is considered to be normal while a score of 20 or higher (indicating at least moderate severity)
HAQ-disability index | Baseline
  There are 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do).The 8 scores of the 8 sections are summed and divided by 8.
SF-36 | Baseline
  Covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Time from first manifestation to diagnosis | Baseline
  Time from first manifestation to diagnosis
Patients prescribed to different treatments | Baseline
  Percentage of patients prescribed to different treatment among naïve and switchers groups; determinants of untreated, treated discontinue, treated persisting status.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pisani, MD, Principal Investigator — Università degli Studi di Napoli "Federico II" NAPOLI; Federico Pieruzzi, MD, Principal Investigator — Ospedale San Gerardo MONZA; Renzo Mignani, MD, Principal Investigator — AUSL della Romagna - Ospedale Infermi RIMINI; Elena Verrecchia, MD, Principal Investigator — Fondazione Policlinico Universitario "Gemelli" IRCCS ROMA; Davide Noto, MD, Principal Investigator — A.O.U. Policlinico "Giaccone" PALERMO; Antonino Tuttolomondo, MD, Principal Investigator — A.O.U. Policlinico "Giaccone" PALERMO; Maurizio Pieroni, MD, Principal Investigator — AUSL Toscana Sud-Est - Ospedale San Donato AREZZO; Iacopo Olivotto, MD, Principal Investigator — A.O.U. Careggi FIRENZE
Locations (7):
- Italy (7):
  - AUSL Toscana Sud-Est - Ospedale San Donato, Arezzo
  - A.O.U. Careggi, Florence
  - U.O.C. Nefrologia ASST Monza - Ospedale San Gerardo, Monza
  - U.O. di Nefrologia - Dipartimento di Sanità Pubblica Università degli Studi di Napoli "Federico II" NAPOLI, Napoli
  - A.O.U. Policlinico "Giaccone", Palermo
  - AUSL della Romagna - Ospedale Infermi, Rimini
  - Fondazione Policlinico Universitario "Gemelli" IRCCS, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CSR Synopsis published on the Chiesi Group web-site — https://www.chiesi.com/en/chiesi-clinical-study-register/